CLINICAL TRIAL: NCT03754777
Title: Evaluation of Modified Enhanced Recovery Program in Emergency Surgery
Brief Title: Modified Enhanced Recovery Program in Emergency Surgery (MERES)
Acronym: MERES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERES
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-09

CONDITIONS: Acute Appendicitis; Acute Appendicitis With Rupture; Acute Appendicitis With Peritonitis; Acute Appendicitis Without Peritonitis
Keywords: enhanced recovery; fast-track; appendectomy; intraperitoneal anesthesia; low pressure pneumoperitoneum
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ERAS protocol group (Experimental): Laparoscopic appendectomy with modified ERAS protocol group Preadmission. Not available due to the emergency setting. Preoperative care.
  1) Patient brochure with a detailed description of the type of pathology, surgery procedure, rehabilitation process, possible complications, and other.
  Surgery.
  1. Low pressure (8-9 mmHg) pneumoperitoneum.
  2. Routinely remove of appendix mesentery in presence of any signs of its inflammation.
  3. Additional local anesthesia with 0.25% ropivacaine.
  4. Abdominal cavity draining only in patients with perforated appendicitis and diffuse peritonitis (Gomes 5).
  Postoperative care.
  1. Early mobilization (2 h after surgery)
  2. Early fluid intake (2 h after surgery)
  3. Early liquid food (6 h after surgery)
  Interventions: Procedure: Laparoscopic appendectomy
- Standard care group (Placebo Comparator): Standard care laparoscopic appendectomy. Preadmission. Not available due to emergency setting. Preoperative care. 1) Patient oral informing about the type of pathology, surgery procedure and possible complications. No brochure.
  Surgery.
  1. Standard pressure (12-14 mmHg) pneumoperitoneum
  2. Abdominal draining for patients with perforated and not perforated appendicitis complicated by abscess, local or diffuse peritonitis (Gomez ≥ 3A).
  3. Appendix mesentery removing in the appearance of its necrotic changes.
  4. No intraabdominal anesthesia. Postoperative care.
  1) Mobilization in 4-6 h after surgery 2) Fluid intake in 6 hours 3) Liquid food intake in 12 hours
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Preoperative care in both arms. Crystalloid isotonic solutions and antibiotic prophylaxis 30 min prior to surgery.
  Surgery. General anesthesia with strict control of fluid therapy and hemodynamic changes during surgery. Appendectomy with the use of monopolar coagulation by experienced surgeons following appendix stump ligation by two Roeder knots.
  Postoperative care. Antibiotics for 3-5 days for patients with complicated appendicitis (Gomez ≥ 3A). The postoperative pain level evaluation in rest by VAS in 0 h (immediately after awakening), 2, 6, 12 and 24 h postop. The postoperative analgesic modality "on demand": Ketorolac 30 mg for patients with VAS pain level ≥ 5 cm. Antiemetics in dyspepsia. No iv infusions postoperatively. Intestinal peristalsis evaluation by auscultation every 2 h after surgery.

SUMMARY:
Laparoscopic appendectomy (LA) is a widespread surgical procedure. Patients may develop considerable postoperative pain and dyspepsia resulting in prolong in-hospital stay. Almost 10% of patients develop postoperative complications. Enhanced recovery after surgery (ERAS) program has proven its effectiveness in elective surgery and can theoretically improve outcomes of LA. To date there is no ERAS program for LA. The aim of the study was to investigate the safety and efficacy of a modified ERAS protocol in LA.

DETAILED DESCRIPTION:
A modified ERAS (mERAS) protocol was investigated. The study is a prospective, randomized nonblinded. All patients underwent LA. Modified ERAS protocol included patient informing, limitation of drainage use; intraperitoneal anesthesia with long-acting anesthetics; low-pressure pneumoperitoneum; early mobilization and oral nutrition. Pain level was assessed in rest using visual analogue scale (VAS). The primary endpoint was postoperative length of stay (pLOS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stage of acute appendicitis except 3B according to Gomes classification;
* Class I-II surgical patients according to the classification of The American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* Patient refusal to participate in the study or to sign the informed consent form;
* Language barrier;
* Transfer to the intensive care unit (ICU) after surgery;
* ASA class ≥ III;
* Conversion to open procedure;
* Appendicular mass found during laparoscopy;
* Gomes 3B appendicitis requiring immersion of the appendicular stump;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay (pLOS) | 30 days
  Time interval measured from the end of the surgery until the moment of discharge from the hospital, measured in days

SECONDARY OUTCOMES:
Complication rate | 30 days
  Number of patients who develop postoperative complications (surgical site infections, intraabdominal organ-specific infection, postoperative ileus) in relation to the total number of patients, measured in percentage
Readmission rate | 30 days
  Number of patients with readmission to the hospital after discharge in relation to the total number of patients, measured as a percentage
Postoperative pain | 24 hours
  Level of postoperative pain syndrome measured with a visual analog scale in centimeters
Shoulder pain incidence | 24 hours
  Quantity of patients who developed shoulder pain after surgery in relation to the total number of patients, measured as a percentage
Shoulder pain level | 24 hours
  Level of shoulder pain syndrome measured with visual analog scale in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Sazhin, Prof., Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Taras Nechay, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sazhin AV, Nechay TV, Titkova SM, Petukhov VA, Tyagunov AE, Stradymov EA, Ermakov IV, Mishakina NY. [Appendectomy technique: paradigm shift or a well-forgotten old one? The role of mesoappendectomy in prevention of infectious intra-abdominal complications (announcement of RCT)]. Khirurgiia (Mosk). 2020;(10):49-59. doi: 10.17116/hirurgia202010149. Russian. PMID 33047586
- [Derived] Nechay T, Sazhin A, Titkova S, Tyagunov A, Anurov M, Melnikov-Makarchuk K, Tyagunov A. Evaluation of enhanced recovery after surgery program components implemented in laparoscopic appendectomy: prospective randomized clinical study. Sci Rep. 2020 Jul 1;10(1):10749. doi: 10.1038/s41598-020-67591-5. PMID 32612104